CLINICAL TRIAL: NCT04413045
Title: Prevalence and Clinical Characteristics of Novel COVID-19 Cases at One Quarantine Hospital; a National Analysis
Brief Title: Novel COVID-19, A National Analysis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed F. Mostafa, Associate Professor of Anesthesia and Intensive Care, Assiut University
Other Study IDs: Novel COVID-19 Prevalence
Record Dates: First submitted 2020-06-01; First posted 2020-06-02 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- C Group: All COVID-19 cases to be admitted in the assigned hospital with positive results of nasopharyngeal swab for SARS-CoV-2 during one-month duration.
  Interventions: Other: Prevalence of COVID-19

INTERVENTIONS:
Other: Prevalence of COVID-19 — All COVID-19 cases to be admitted in the assigned hospital with positive results of nasopharyngeal swab for SARS-CoV-2 during one-month duration.

SUMMARY:
Pneumonia is a form of acute respiratory tract infection (ARTI) that affects the lungs. When an individual has pneumonia, the alveoli in the lungs are filled with pus and fluid, which makes breathing painful and limits oxygen intake. Pneumonia has many possible causes, but the most common are bacteria and viruses but nowadays there is a pandemic spread from novel corona virus which cause corona virus disease 2019 (COVID-19).

Corona virus comprises of a large family of viruses that are common in human beings as well animals (camels, cattle, cats, and bats). There are seven different strains of corona virus. Sometimes corona virus from animals infect people and spread further via human to human transmission such as with MERS-CoV, SARS-CoV, and now with this COVID-19 (Corona disease 2019). The virus that causes COVID-19 is designated as severe acute respiratory syndrome corona virus 2 (SARS-CoV-2); previously, referred to as 2019-nCoV.

On Towards December 2019, this novel corona virus was identified as a cause of upper and lower respiratory tract infections in Wuhan, a city in the Hubei Province of China. It rapidly spread, resulting in an epidemic throughout China and then gradually spreading to other parts of the world in pandemic proportions. It has affected almost every continent in this world. In February 2020, the World Health Organization designated the disease COVID-19, which stands for corona virus disease 2019.

The Coronaviruses are a large family of single-stranded RNA viruses (+ssRNA) that can be isolated in different animal species. They have a crown-like appearance under an electron microscope (coronam is the Latin term for crown) due to the presence of spike glycoproteins on the envelope. These viruses can also infect humans and cause illness ranging from the common cold to more severe diseases such as MERS, SARS and now COVID-19. According to recent research, a spike mutation, which probably occurred in late November 2019, triggered jumping to humans.

DETAILED DESCRIPTION:
This study will be done at one quarantine hospital in Assiut, Egypt. After approval from our Institutional Ethics Committee, a written informed consent will be obtained from all patients or their legal representatives (if they are unable to provide consent) before enrollment in the study.

Study Design and Sample Size Calculation: This study is an investigator-initiated cross sectional trial to record, assess the clinical manifestations and prognosis of all COVID-19 cases to be admitted in the assigned hospital with positive results of nasopharyngeal swab for SARS-CoV-2 during one-month duration. According to our records, 30-60 patients may be included.

Clinical Classification of COVID-19 patients according to the Egyptian Ministry of Health and Population:

* Mild Cases: The clinical symptoms are mild and no pneumonia manifestations can be found in imaging.
* Moderate Cases Patients have symptoms (such as fever and respiratory tract symptoms, etc.) and pneumonia manifestations can be seen in imaging.
* Severe Cases Adults who meet any of the following criteria: Respiratory rate< 30 breaths/min; Oxygen saturations < 93% at a rest state; Arterial partial pressure of oxygen (PaO2)/Fraction of inspired oxygen (FiO2) [P/F ratio] <300 mmHg; Patients with more than 50% lesions progression within 24 to 48 hours in lung imaging should be treated as severe cases.

Study Tools and Data Collection: All admitted patients to the hospital will be monitored carefully and observed for medical treatment, supportive measures, hemodynamic variables, and comorbid conditions.

* Demographic Data: including age, sex and occupation.
* History of travelling abroad and history of contact to confirmed cases (positive to SARS-CoV-2).
* Vital signs (heart rate, non-invasive blood pressure, respiratory rate, peripheral oxygen saturation) at admission, at day 3, and day 7.
* laboratory investigation:

  * Complete blood picture
  * CRP (C reactive protein)
  * Prothrombin time, concentration, and INR
  * Liver function (ALT, AST, bilirubin)
  * Kidney function (blood urea and serum creatinine)
  * Arterial blood gas (ABG): at admission, day1, day 3 and day 5.
  * D-Dimer and ferritin levels
  * HRCT chest (High resolution computed tomography) chest at admission and follow up at discharge.
* Follow up and outcome: (RT-PCR for SARS-CoV-2, CT chest, ABG).
* The need of invasive mechanical ventilation, the clinical outcome, the duration of ICU and hospital stay.
* Any complications

ELIGIBILITY:
Inclusion Criteria:

* Any Age
* Any Sex
* non pregnant women
* RT-PCR positive for SARS-CoV-2

Exclusion Criteria:

* Patient Refusal
* Pregnancy
* patients stopped participation at anytime

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is an investigator-initiated cross sectional trial to record, assess the clinical manifestations and prognosis of all COVID-19 cases to be admitted in the assigned hospital with positive results of nasopharyngeal swab for SARS-CoV-2 during one-month duration.
  The study aims To detect epidemiology, clinical and radiological presentation, laboratory findings, complications, duration needed to conversion from positive to negative PCR, duration of hospital stay and outcome of COVID-19 patients admitted in one quarantine hospital
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Patient Prognosis Score | 1 month
  The prognosis of COVID-19 patients at one quarantine hospital delivered to home, prolonged hospital stay, death.

SECONDARY OUTCOMES:
Oxygen Saturation | 14 days
  Non-invasive peripheral oxygen saturation (%)
Laboratory Data | 14 days
  Complete blood picture
Radiological Features | 1 month
  High resolution computed tomography chest at admission and follow up at discharge
Hospital Stay | 1 month
  Duration of patients stay at hospital
Liver Function | 1 month
  Complete liver function tests
Kidney Function | 1 month
  Complete liver function tests

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F. Mostafa, MD, Principal Investigator — membership/educator
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided